CLINICAL TRIAL: NCT07387809
Title: Clinical Investigation of the Effectiveness of Laser-activated Photoacoustic Flow in One-visit Revision of Teeth With Apical Periodontitis
Brief Title: Effectiveness of Laser-activated Photoacoustic Flow in One-visit Revision of Teeth With Apical Periodontitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Domagoj Kunčić, Dr. Domagoj Kunčić, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-PA-2-5/2025; School of Dental Medicine (Other: University of Zagreb)
Record Dates: First submitted 2026-01-01; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Apical Periodontitis
Keywords: apical periodontitis; laser-activated irrigation; single-visit revision
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSP modality of Er:YAG laser activated irrigation (Experimental): In group 1, irrigant in the final irrigation protocol will be activated by a radial laser attachment (diameter: 400 µm) of an Er:YAG laser (Fotona, Ljubljana, Slovenia). The laser settings will be: SSP mode, pulse energy 20 mJ, frequency 15 Hz, pulse duration 50 µs according to the factory settings of the Er:YAG laser for laser-activated disinfection and according to the endodontic space disinfection protocol (23).
  Interventions: Device: Laser activated irrigation
- Sound-activated irrigation (Smart Lite Pro EndoActivator, DentsplySirona) (Active Comparator): In group 2, each irrigant in the final irrigation protocol will be activated by the polymer tip of the sonic irrigation device. The tip will be placed 2 mm from the working length of the canal. The activation time will be 30 s for NaOCL, 60 s for EDTA and 30 s for NaOCl.
  Interventions: Device: Sound-activated irrigation

INTERVENTIONS:
Device: Laser activated irrigation — In this group, the final irrigation protocol will be activated by an Er:YAG laser (Fotona, Ljubljana, Slovenia) in SSP mode.
  Arms: SSP modality of Er:YAG laser activated irrigation
Device: Sound-activated irrigation — In this group, the final irrigation protocol will be activated by the polymer tip of the sonic irrigation device.
  Arms: Sound-activated irrigation (Smart Lite Pro EndoActivator, DentsplySirona)

SUMMARY:
The main objective of the clinical randomized study is to examine the effectiveness laser-activated irrigation (LAI) on the removal of intracanal microorganisms and the healing of an inflammatory periapical lesion of a tooth after a one-visit revision of teeth with apical periodontitis.

The main questions are:

1. Does LAI reduces the occurrence of postoperative pain, compared with sonic-activated irrigation?
2. Is antimicrobial efficacy of LAI greater than the antimicrobial efficacy of sonic-activated irrigation?
3. Is periapical lesion healing after LAI application better than after sonic-activated irrigation?

Researcher will compare LAI and sonic-activated irrigation in patients with signs and symptoms of chronic apical periodontitis requiring revision. Participants will be assigned to two experimental groups depending on the final root canal disinfection protocol. Postoperative pain will be assessed via a questionnaire that participants will receive after the treatment and which they will complete over a period of seven days. Microbiological samples will be collected from the root canal and real-time PCR analysis will be performed to evaluate antimicrobial efficacy. Assessment of periapical lesion healing will be performed by comparing CBCT scans obtained before the treatment and one year after.

DETAILED DESCRIPTION:
Introduction:

Endodontic treatment of teeth involves thorough mechanical removal of microorganisms, necrotic and infected pulp tissue, and chemical disinfection of the endodontic space. Due to the complex morphology of the endodontic space, which includes lateral canals, isthmuses, and apical bifurcations, more than a third of the root canal remains untreated after mechanical treatment, so chemical disinfection is an indispensable addition to mechanical treatment. The work of instruments in the root canal creates a residual layer on the canal walls, and dentin debris created by instrumentation accumulates in the irregularities of the canal and serves as an ideal refuge for remaining bacteria. In addition, the residual layer on the dentin walls can prevent the penetration of irrigant and filler into the dentinal tubules. Therefore, abundant irrigation with irrigant is essential for removing dentin chips from the root canal, but also the residual layer from its walls.

Ultrasonic and laser-activated disinfection are increasingly used to improve the depth of penetration of the irrigant used and thus reduce persistent periradicular inflammation. However a systematic review from 2023 that laser-activated disinfection is significantly better at reducing the number of microorganisms and removing residual layer and dentine debris compared to ultrasonically activated disinfection. It is believed that laser-activated disinfection improves the effectiveness of irrigant in disinfecting the endodontic space by creating secondary cavitations through expansion and subsequent implosion of the liquid. Er:YAG lasers use laser energy to create acoustic waves that move the irrigant and thus improve its flow inside the root canal, which is especially true for the PIPS technique (photon-induced photoacoustic streaming). It is shown that laser-activated disinfection, in vitro, can reduce the number of bacteria in infected canals by 99.5%. Modalities of the Er:YAG laser, such as SWEEPS (shock wave enhanced emission photoacoustic streaming) and SSP (super short pulse), create a precise concentration of shock waves during irrigation, which enable the washing agent to penetrate deeper into the lateral canals and microscopic tubules, thereby increasing the effectiveness of disinfection. Because of the above, SWEEPS/SSP modalities have significant advantages during endodontic treatment, especially in teeth with complicated root canal morphology.

However, although in vitro studies show that laser-activated irrigation (LAI) is superior to other methods in removing intracanal microorganisms, there are still very few clinical studies. Clinical studies show that the healing of periapical lesions after one year on single-rooted teeth and premolars is the same for all irrigation techniques. However, a higher percentage of healing has also been reported when using the SWEEPS modality. It is also emphasized the need for additional research that would study the effectiveness of LAI in multi-rooted teeth, considering their more pronounced morphology of the endodontic space, on which pulsed laser modalities could be more effective.

There is also increasing emphasis on the use of cone-beam computed tomography (CBCT) in future studies to assess prognostic factors affecting the outcome of root canal treatment. Periapical radiographs show a more favorable outcome of healing of periapical lesions compared to CBCT, which significantly affects the correct assessment of treatment success. The ESE guidelines recommend clinical and radiographic follow-up for at least one year after endodontic treatment, with the patient's radiation dose as low as possible to achieve the desired level of diagnosis. The use of CBCT with ethical approval is justified in the clinical use of small CBCT scans for research purposes: to evaluate treatment with new protocols, disinfection techniques, which will provide a more objective treatment outcome.

Furthermore, in addition to the evaluation of LAI on the healing of periapical lesions, one of the important issues is the impact of LAI on postoperative pain. Namely, during endodontic procedures, a major problem encountered is postendodontic pain, which, with its incidence of 3-58%, is a relatively common occurrence. Although it has been reported that LAI results in lower levels of postoperative pain, the number of clinical studies is small, and they show conflicting results on whether LAI is superior to other techniques. However, studies which did not find a difference in LAI and ultrasonic irrigation only investigated asymptomatic lesions in primary endodontic treatment. In contrast, it was reportoed that postoperative pain is significantly less intense when LAI is used compared to other techniques in the treatment of symptomatic irreversible pulpitis. Likewise, a recent meta-analysis showed that pulsed Er:YAG modalities, especially SWEEPS, have a stronger analgesic effect compared to ultrasound irrigation.

Given that the long-term goal of endodontic therapy is to maintain the masticatory and aesthetic function of the teeth, the goal of this study was to determine the effectiveness of laser-activated root canal disinfection during a one-visit revision of the treatment of teeth with apical periodontitis.

Objectives:

The main objective of the clinical randomized study is to examine the effectiveness of the Super Short Pulse (SSP) modality of Er:YAG laser-activated irrigation (LAI) on the removal of intracanal microorganisms and the healing of an inflammatory periapical lesion of a tooth after a one-visit revision.

Secondary objective:

1. To examine the effect of the Super Short Pulse (SSP) modality of Er:YAG laser-triggered lavage applied during a single-visit revision, on the occurrence of postoperative pain, compared with sound-triggered lavage.
2. To compare the antimicrobial efficacy of SSP ER:YAG LAI with the antimicrobial efficacy of sound-activated rinsing
3. To compare the healing of the periapical lesion after the application of SSP ER:YAG LAI during a one-visit revision of the tooth with the healing of the lesions after the application of sound-activated irrigation

Matherials and methods:

A randomized clinical trial will be conducted at the Department of Endodontics and Restorative Dental Medicine, School of Dental Medicine, University of Zagreb (Gundulićeva 5). All procedures in conducting the study were approved by the Ethics Committee of the School of Dental Medicine, University of Zagreb (Approval Number: 05-PA-2-5/2025; Date: 17 February 2025) and are in accordance with the Declaration of Helsinki.

Participants Patients with signs and symptoms of chronic apical periodontitis requiring revision will be included in the study. The diagnosis will be determined based on the history, clinical examination, and X-ray analysis.

Inclusion criteria: teeth tender to percussion, palpation, teeth that have a sinus tract and swelling, a chronic periapical lesion greater than 5 mm in diameter based on the initial X-ray (which the patient brings at the first examination) and previous endodontic treatment and root canal filling that is inadequate according to clinical criteria (filling, overfilling, non-homogeneous root canal filling, unfilled root canals).

Exclusion criteria: immunocompromised patients, pregnant women, teeth with a periodontal pocket depth greater than 3 mm, teeth with signs and symptoms of vertical fracture, teeth that cannot be restored or prosthetically provided after endodontic treatment, use of antibiotic therapy within the last month, and diagnosis of acute apical abscess.

All respondents included in the study will sign an informed consent form for the use of personal data and will receive written information about the study. All respondents will be able to withdraw from the study at any time during the study.

Before the start of the endodontic treatment, each subject will be randomly assigned to one of two experimental groups. Randomization will be performed based on the WheelDecide program (www.wheeldecide.com). All phases of endodontic treatment of teeth will be performed by a doctoral student with more than five years of experience in endodontic treatment of teeth. All subjects will undergo a single-visit endodontic treatment of teeth. Subjects will be assigned to two experimental groups depending on the final root canal disinfection protocol. In both groups, the final irrigation protocol will include the following standard sequence of irrigant: 1) 3% sodium hypochlorite (NaOCl), 2) ethylenediaminetetraacetic acid (EDTA), and 3) 3% NaOCl.

Group 1. SSP modality of Er:YAG laser activated irrigation In group 1, each irrigant in the final irrigation protocol will be activated by a radial laser attachment (diameter: 400 µm) of an Er:YAG laser (Fotona, Ljubljana, Slovenia). The laser settings will be: SSP mode, pulse energy 20 mJ, frequency 15 Hz, pulse duration 50 µs according to the factory settings of the Er:YAG laser for laser-activated disinfection and according to the endodontic space disinfection protocol (15).

Group 2. sound-activated irrigation (Smart Lite Pro EndoActivator, DentsplySirona) In group 2, each irrigant in the final irrigation protocol will be activated by the polymer tip of the sonic irrigation device. The tip will be placed 2 mm from the working length of the canal. The activation time will be 30 s for NaOCL, 60 s for EDTA and 30 s for NaOCl.

The endodontic procedure in all subjects will be performed according to modern endodontic treatment guidelines. The endodontic procedure will be performed under local (conduction or infiltration) anesthesia (articaine 4% with adrenaline in a ratio of 1:100,000) and rubber dam isolation. In all subjects, the treatment procedure will be performed with the ProTaperNext rotary system (DentsplySirona, Germany) with mechanical canal treatment instruments with motor settings: 300 rpm and 300 Ncmtorque. The initial working length will be determined with hand instruments: K-file #10 or #15 to the apical foramen (value 0 on the apex locator). During mechanical canal preparation, the canals will be irrigated with a total of 5 ml of 3% NaOCl per canal with 30G SteriTips side vented needles, which will be placed approximately 4 mm from the working length.

After the chemo-mechanical treatment of the canals, a final disinfection protocol will be carried out for each patient, depending on which group they belong to. In each group, the canals will be filled with a calcium silicate-based filler (BioRoot RCS, Septodont, Saint-Maur-des-Fossés Cedex, France) using a single gutta-percha stick technique. All teeth will be temporarily closed with glass ionomer cement (Equia Forte, GC, Tokyo, Japan). At the next visit, a permanent composite filling will be placed.

Microbiological sampling and analysis

Microbiological samples will be collected from the root canal:

Sample 1. After trepanation of the tooth Sample 2. After chemo-mechanical canal preparation Sample 3. After final irrigation protocol Strict aseptic conditions will be applied for sample collection during endodontic treatment. The paper swab with which the sample was collected will be placed in a cryochamber containing Tris-EDTA buffer (10 mmol/L Tris-HCl, 1 mmol/L EDTA, pH = 7.6) and immediately frozen at -20 degrees Celsius. Real-time PCR analysis will be performed.

Quantitative analysis of periapical lesion healing on CBCT images Before the start of endodontic treatment, an initial CBCT image of the target tooth will be made in all patients for the purpose of initial diagnosis, analysis of the anatomy of the endodontic space and assessment of the extent of the periapical lesion, based on which a decision will be made on the therapeutic procedure: endodontic treatment, revision or tooth extraction. The application of CBCT will be carried out according to the guidelines of the European Society of Endodontics. All CBCT images will be made on the same CBCT device with the same imaging parameters (endomod, voxel size 0.085 mm, 450.3 mGy/cm2, 6.3mA, 90kV, 8.7s). All radiation doses to the subjects will be "as low as reasonably achievable" (ALARA).

In order to assess the long-term prognosis of the tooth and decide on future prosthetic or surgical therapy, a control CBCT will be made 12 months later, according to the same parameters as in the first scan.

The healing analysis will be performed by two experienced endodontists with prior calibration. Each endodontist will place each scanned tooth in a specific category according to the following criteria.

1. New periapical radiolucency
2. Increased periapical radiolucency
3. Unchanged periapical radiolucency
4. Reduced periapical radiolucency according to which a decision will be made on further procedures: endodontic surgery, tooth monitoring, tooth extraction. Any disagreement in the decision will be resolved by discussion until an agreement is reached.

The healing analysis of the lesion will be performed by volumetric assessment using the ITK-SNAP software. Calculation and volumetric assessment in mm3 will be performed with ITK-SNAP with additional shaping, manual adjustment and transfer. In multi-rooted teeth, the defect will be displayed as the sum of individual periapical processes. At the 12-month check-up, all processes smaller than twice the thickness of the periodontal ligament will be counted as 0 mm3, or complete healing.

Postoperative pain assessment after a single-visit dental revision After the procedure, the subjects will receive a questionnaire on the occurrence, duration and intensity of postoperative pain, which they will fill out over a period of seven days.

Statistical procedures The Chi-square test, Fisher's exact test and Fisher-Freeman-Halton test will be used for statistical analysis. The significance level will be set at 5%. The tests for postoperative pain were the percussion test and the palpation test.

ELIGIBILITY:
Inclusion Criteria:

* teeth tender to percussion, palpation
* teeth that have a sinus tract and swelling
* a chronic periapical lesion greater than 5 mm in diameter based on the initial X-ray
* previous endodontic treatment and root canal filling that is inadequate according to clinical criteria (filling, overfilling, non-homogeneous root canal filling, unfilled root canals)

Exclusion Criteria:

* immunocompromised patients
* pregnant women
* teeth with a periodontal pocket depth greater than 3 mm
* teeth with signs and symptoms of vertical fracture
* teeth that cannot be restored or prosthetically provided after endodontic treatment
* use of antibiotic therapy within the last month
* diagnosis of acute apical abscess

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | From day 1 after treatment to 7 days postoperatively
  Following single-visit revision performed with different irrigation activation techniques, occurance, duration and intensity of postoperative pain will be assessed via a questionnaire. A score of 0 represented no pain, while a score of 10 represented the maximum pain, with higher scores indicating greater pain intensity.
Radiographic healing of periapical lesions | At the 12-month
  The healing analysis of the lesion will be performed by volumetric assessment using the ITK-SNAP software. Calculation and volumetric assessment in mm3 will be performed with ITK-SNAP with additional shaping, manual adjustment and transfer. In multi-rooted teeth, the defect will be displayed as the sum of individual periapical processes. All processes smaller than twice the thickness of the periodontal ligament will be counted as 0 mm3, or complete healing.

SECONDARY OUTCOMES:
Microbiological efficiency | At the baseline
  Real-time PCR analysis will be performed to determine bacteria quantity. Samples from the root canal will be collected at the time of first appointment during single visit revision in 3 stages of procedure: 1. after trepanation; 2. after chemo-mechanical preparation and 3. after final irrigation protocol

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dental Medicine, University of Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Davies A, Mannocci F, Mitchell P, Andiappan M, Patel S. The detection of periapical pathoses in root filled teeth using single and parallax periapical radiographs versus cone beam computed tomography - a clinical study. Int Endod J.2015;48(6):582-92.
- [Background] Sabeti M, Harouni A, Gabbay J. Comparing Ultrasonically Activated Irrigation and Laser-Activated Irrigation for Postoperative Pain Reduction in Endodontics: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Endod. 2026 Jan;52(1):37-46.
- [Background] Erkan E, Gündoğar M, Uslu G, Özyürek T. Postoperative pain after SWEEPS, PIPS, sonic and ultrasonic-assisted irrigation activation techniques: a randomized clinical trial. Odontology. 2022 Oct;110(4):786-794.
- [Background] Liapis D, De Bruyne MAA, De Moor RJG, Meire MA. Postoperative pain after ultrasonically and laser-activated irrigation during root canal treatment: a randomized clinical trial. Int Endod J. 2021 Jul;54(7):1037-1050.
- [Background] Sathorn C, Parashos P, Messer H. The prevalence of postoperative pain and flare- up in single- and multiple- visit endodontic treatment: a systematic review. Int Endod J. 2008;41 (2)91-99.
- [Background] Duncan HF, Kirkevang LL, Peters OA, El-Karim I, Krastl G, Del Fabbro M, Chong BS, Galler KM, Segura-Egea JJ, Kebschull M; ESE Workshop Participants and Methodological Consultant. Treatment of pulpal and apical disease: The European Society of Endodontology (ESE) S3-level clinicalpracticeguideline. Int Endod J. 2023 Oct;56 Suppl 3:238-295.
- [Background] Davies A, Patel S, Foschi F, Andiappan M, Mitchell PJ, Mannocci F. The detection of periapical pathoses using digital periapical radiography and cone beam computed tomography in endodontically retreated teeth - part 2: a 1 year post-treatment follow-up. Int Endod J. 2016;49:623-35;
- [Background] Patel S, Wilson R, Dawood A, Mannocci F. The detection of periapical pathosis using periapical radiography and cone beam computed tomography - part 1: preoperative status. Int Endod J. 2012;45:702-10.
- [Background] Doğan MU, Arıcıoğlu B, Köse TE, Çıkman AŞ, Öksüzer MÇ. Association between the irrigation-agitation techniques and Periapical Healing of large periapical lesions: a Randomized Controlled Trial. Clin Oral Investig. 2024 Jun 15;28(7):376.
- [Background] Martins MR, Carvalho MF, Pina-Vaz I, Capelas JA, Martins MA, Gutknecht N. Outcome of Er,Cr:YSGG laser-assisted treatment of teeth with apical periodontitis: a blind randomized clinical trial. Photomed Laser Surg. 2014 Jan;32(1):3-9.
- [Background] Josic U, Mazzitelli C, Maravic T, Fidler A, Breschi L and Mazzoni A. Biofilm in endodontics: in vitro cultivation possibilities, sonic-, ultrasonic- and laser-assisted removal techniques and evaluation of the cleaning efficacy. Polymers (Basel), 2022;14, 1334.
- [Background] Do QL, Gaudin, A. The efficiency of the Er: YAG laser and photoninduced photoacoustic streaming (PIPS) as an activation method in endodontic irrigation: a literature review. JLMS. 2020;11,316-334.
- [Background] Jordana J, Tandean JN, Salim JF, Jennifer, Febriastuti C, Sampoerno G. Shock wave enhanced emission photoacoustic streaming (SWEEPS): An alternative to conventional irrigation in endodontic treatment. Conservative Dentistry Journal. 20122. 12:68-72.
- [Background] Blanken J, De Moor RJ, Meire M, etal. Laser induced explosive vapor and cavitation resulting in effective irrigation of the root canal. Part 1: a visualization study, LasersSurg Med. 2009;41:7.
- [Background] Peters OA, Bardsley S, Fong J, Pandher G, Divito E: Disinfection of root canals with photon-initiated photoacoustic streaming. J.Endod. 2011;1, 37:1008-12.
- [Background] Badami V, Akarapu S, Kethineni H, Mittapalli SP, Bala KR, Fatima SR. Efficacy of Laser-Activated Irrigation Versus Ultrasonic-Activated Irrigation: A SystematicReview. Cureus. 2023;15(3): e36352.
- [Background] Haapasalo M, Shen Y, Wang Z, Gao Y.Irrigation in endodontics. Braz.Dent. J. 2014;216, 299-303.
- [Background] Baumgartner JC, Mader CL. A scanning electronmicroscopic evaluation off our root canal irrigation regimens. J Endod. 1987;13:147-57.
- [Background] McComb D, Smith DC. A preliminary scanning electronmicroscopic study of root canals after endodontic procedures. JEndod. 1975;1, 238-42.
- [Background] Vertucci FJ. Root canal morphology and its relationship to endodontic procedures. Endod Top. 2005;10(1):3-29.